CLINICAL TRIAL: NCT04019808
Title: Interventional Study at the Primary and Secondary Levels of Prevention for Knowledge Regarding GC Risk Factors in EU and CELAC Populations
Brief Title: Gastric Cancer Risk Factors Knowledge in European and Latinamerican Population
Acronym: LEGACY-3
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: Instituto Nacional de Cancerologia de Mexico (Other); Amsterdam UMC, location VUmc (Other); Pontificia Universidad Catolica de Chile (Other); Vall d'Hebron Institute of Oncology (Other); INSTITUTO ALEXANDER FLEMING (Unknown); Hospital Central del IPS (Other); IPATIMUP - Instituto De Patologia E Imunologia Molecular Da Universidade Do Porto (Other)
Responsible Party: Sponsor
Other Study IDs: LEGACY-3
Record Dates: First submitted 2019-06-05; First posted 2019-07-15 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Personalized medicine; Oncology; Solid tumor; Primary Intervention
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is divided into two parts:

Part 1: An interventional study, with a pre-post study design to determinate the grade of knowledge of established GC risk factors.

Part 2: An observational study to know impact on prevalence and infection eradication of H. pylori

DETAILED DESCRIPTION:
Part 1: to determinate the grade of knowledge of established GC risk factors and identification of attitudes about, GC screening programs at baseline, prior to the intervention though an educational program.

Part 2: to generate an H. pylori registry, to know its impact on prevalence and infection eradication rate at 6th, 12th, 24th and at Month 36th.

ELIGIBILITY:
Part A: Educational Intervention Inclusion criteria

* Subjects >18 years old, from EU and CELAC countries participating in this study.
* Has given and signed the IC to participate in this study. Exclusion criteria
* Subjects who have received some prior preparation (Cancer Gastric Information).
* Subjects who have previous Knowledge in Gastric Cancer (Example, near relatives who have suffered Gastric Cancer

Part B: H. pylori Register Inclusion criteria

* Subjects ≥18 years old diagnose from H. pylori infection and treated at participant sites
* Has given and signed the IC. Exclusion criteria
* Subjects with chronic gastritis without confirmed diagnose of H. pylori infection, pathologically of by urease test.
* Patient's with CG diagnosis (including gastroesophageal junction cancer).

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Part 1:
  Subjects >18 years old whom able to answer the questions structured in the survey.
  Part 2:
  Subjects >18 years old diagnose from H. pylori infection
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
knowledge GC risk factors and symptoms | 3 years
  Compare the results obtained through a knowledge of CG risk factors by study-specific questionnaire before and after an educational intervention
H. pylori prevalence and drug resistance | 3 years
  Generate an H. pylori registry, to know its impact on prevalence and infection eradication rate at months 6th, 12th, 24th and 36th.

CONTACTS AND LOCATIONS:
Locations (8):
- Instituto Alexander Fleming, Buenos Aires, Argentina
- Pontificia Universidad Católica de Chile, Santiago, Chile
- Instituto Nacional de Cancerología, México, Mexico
- VU Medical Centre, Amsterdam, Netherlands
- GenPat, Asunción, Paraguay
- Institute of Pathology and Immunology of University of Porto, Porto, Portugal
- Spain (2):
  - Fundació Privada Institut d'Investigació Oncològica de Vall-Hebron (VHIO), Barcelona
  - Fundación Investigación Clínico de Valencia, Valencia

REFERENCES:
- [Derived] Carbonell-Asins JA, Jimenez-Marti E, Romero S, Garcia E, Miralles-Marco A, Lopez B, Huerta M, Caballero C, Boggino H, Gauna C, Acevedo-Funes OB, Nunez GB, Cespedes-Cardozo CM, Fernandez-Figueroa EA, Ortiz-Olvera N, Ruiz-Garcia E, Carneiro F, Barros R, Figueiredo C, Ferreira RM, Groen-van Schooten TS, van Santvliet D, Derks S, Luca R, Alsina M, Riquelme A, Cervantes A, Fleitas T. Implementation of an Educational Intervention for Gastric Cancer Awareness in the General Population in CELAC and Europe: A Strategy Proposed by the LEGACy Consortium. J Cancer Educ. 2025 Oct;40(5):804-811. doi: 10.1007/s13187-025-02578-2. Epub 2025 Feb 13. PMID 39939517
- [Derived] van Schooten TS, Derks S, Jimenez-Marti E, Carneiro F, Figueiredo C, Ruiz E, Alsina M, Molero C, Garrido M, Riquelme A, Caballero C, Lezcano E, O'Connor JM, Esteso F, Farres J, Mas JM, Lordick F, Vogt J, Cardone A, Girvalaki C, Cervantes A, Fleitas T; members of LEGACy consortium. The LEGACy study: a European and Latin American consortium to identify risk factors and molecular phenotypes in gastric cancer to improve prevention strategies and personalized clinical decision making globally. BMC Cancer. 2022 Jun 13;22(1):646. doi: 10.1186/s12885-022-09689-9. PMID 35692051